CLINICAL TRIAL: NCT03402243
Title: Effect of Banning Menthol Flavorant on Cigarette and E-Cigarette Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R03DA045150 (NIH); R03DA045150 (NIH)
Record Dates: First submitted 2018-01-09; First posted 2018-01-18 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Menthol ban only for cigarettes (Experimental): Participants will have available to them non-menthol cigarettes, menthol and tobacco flavored versions of a cigarette-like e-cigarette, menthol and tobacco flavored versions of a tank like e-cigarette and nicotine gum and lozenge
  Interventions: Other: Menthol ban on cigarettes
- Menthol ban for cigarettes and e-cigarettes (Experimental): Participants will have available to them non-menthol cigarettes, tobacco flavored version of a cigarette-like e-cigarette, tobacco flavored version of a tank like e-cigarette and nicotine gum and lozenge
  Interventions: Other: Menthol ban on cigarettes and e-cigarettes
- No Menthol Ban (Other): Participants will have available to them menthol and non-menthol cigarettes, menthol and tobacco flavored versions of a cigarette-like e-cigarette, menthol and tobacco flavored versions of a tank like e-cigarette and nicotine gum and lozenge
  Interventions: Other: No menthol ban

INTERVENTIONS:
Other: Menthol ban on cigarettes — Participants will have menthol and tobacco flavored e-cigarettes available but only non-menthol cigarettes
  Arms: Menthol ban only for cigarettes
Other: Menthol ban on cigarettes and e-cigarettes — Participants will have neither menthol flavored cigarettes or e-cigarettes available
  Arms: Menthol ban for cigarettes and e-cigarettes
Other: No menthol ban — Participant will have menthol and tobacco flavored cigarettes and e-cigarettes available
  Arms: No Menthol Ban

SUMMARY:
In this pilot study, menthol cigarette smokers will be randomized to one of three experimental marketplaces: 1) a condition simulating a ban on menthol cigarettes but not menthol e-cigarettes (condition A); 2) a condition simulating a ban on both menthol cigarettes and menthol e-cigarettes (Condition B); and 3) a condition in which menthol is not banned for either product (Condition C - the control condition). All conditions would have medicinal nicotine available if subjects decide to quit tobacco products entirely. At visits occurring every two weeks over a 6 week period, subjects will receive "credits" that they could exchange for any product available in their randomized marketplace condition. Outcomes include the amount of each tobacco product used.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 64
* Purchase exclusively menthol cigarettes
* Not currently motivated to quit smoking
* Smoking a minimum number of cigarettes per day

Exclusion Criteria:

* Report a serious, unstable medical or psychiatric condition
* Use any medications that might interfere with measures to be studied (for example, medications known to affect smoking)
* Have used any smoking cessation therapy during the past month
* Regularly use any form of tobacco other than cigarettes
* Are pregnant or breast feeding or planning to become pregnant or breast feed during the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Sciences Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable information will be shared with other researchers

REFERENCES:
- [Derived] Kotlyar M, Shanley R, Dufresne SR, Corcoran GA, Hatsukami DK. Effect on Tobacco Use and Subjective Measures of Including E-cigarettes in a Simulated Ban of Menthol in Combustible Cigarettes. Nicotine Tob Res. 2022 Aug 6;24(9):1448-1457. doi: 10.1093/ntr/ntac107. PMID 35430631

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Menthol Ban Only for Cigarettes | Menthol Ban for Cigarettes and E-cigarettes | No Menthol Ban
Started (Number of participants who were informed of their randomization and contributed to the analysis) | 16 | 15 | 16
Completed | 13 | 12 | 14
Not Completed | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menthol Ban Only for Cigarettes | Menthol Ban for Cigarettes and E-cigarettes | No Menthol Ban | Total
Number analyzed (Participants) | 16 | 15 | 16 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (9.8) | 44.9 (11.2) | 44.1 (10.4) | 44.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 9 | 25
  Male | 8 | 7 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 14 | 15 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 5 | 16
  White | 7 | 10 | 9 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Amount of Tobacco Product Used
Description: Total number of cigarettes smoked and puffs of e-cigarettes used
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: tobacco products use per day
Arm/Group | Menthol Ban Only for Cigarettes | Menthol Ban for Cigarettes and E-cigarettes | No Menthol Ban
Number analyzed (Participants) | 16 | 15 | 16
tobacco products use per day
  Cigarettes smoked per day | 13.1 (5.5) | 18.6 (5.7) | 15.3 (5.0)
  Puffs of e-cigarettes used per day | 56.7 (180.2) | 10.7 (24.9) | 4.5 (8.6)
Statistical Analysis 1: Comparison: Menthol Ban Only for Cigarettes vs Menthol Ban for Cigarettes and E-cigarettes; Test type: Superiority; Estimated mean ratio = 1.38, 95% CI 2-sided [1.1 to 1.75] — Baseline adjusted model estimated mean ratio in cigarettes smoked per day of those randomized to a total menthol ban smoked relative to those randomized to a menthol cigarette ban
Statistical Analysis 2: Comparison: Menthol Ban Only for Cigarettes vs No Menthol Ban; Test type: Superiority; Estimated mean ratio = 0.87, 95% CI 2-sided [0.68 to 1.11] — Baseline adjusted model estimated mean ratio in cigarettes smoked per day of those randomized to a menthol cigarettes ban relative to those randomized to no menthol ban
Statistical Analysis 3: Comparison: Menthol Ban for Cigarettes and E-cigarettes vs No Menthol Ban; Test type: Superiority; Estimated mean ratio = 1.20, 95% CI 2-sided [0.99 to 1.45] — Baseline adjusted model estimated mean ratio in cigarettes smoked per day of those randomized to a menthol ban for cigarettes and e-cigarettes relative to those randomized to no menthol ban
Statistical Analysis 4: Comparison: Menthol Ban Only for Cigarettes vs Menthol Ban for Cigarettes and E-cigarettes vs No Menthol Ban; Average number of puffs per participants over the 6 week study period; Test type: Superiority; p = 0.349, Kruskal-Wallis

2. Secondary Outcome: How Much of Each Product is Obtained From the "Experimental Marketplace"
Description: Number of packs of cigarettes obtained and amount of e-liquid obtained from the "experimental marketplace"
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units of tobacco
Arm/Group | Menthol Ban Only for Cigarettes | Menthol Ban for Cigarettes and E-cigarettes | No Menthol Ban
Number analyzed (Participants) | 16 | 15 | 16
units of tobacco
  Packs of cigarettes | 22.6 (10.38) | 29.3 (11.06) | 28.8 (10.7)
  Units of e-cigarette liquid | 3.13 (3.16) | 1.2 (1.57) | 1.06 (1.34)
Statistical Analysis 1: Comparison: Menthol Ban Only for Cigarettes vs Menthol Ban for Cigarettes and E-cigarettes vs No Menthol Ban; Comparison among groups in number of cigarette packs selected; Test type: Superiority; p = 0.185, Mixed Models Analysis
Statistical Analysis 2: Comparison: Menthol Ban Only for Cigarettes vs Menthol Ban for Cigarettes and E-cigarettes vs No Menthol Ban; Comparison among groups in number of e-cigarette liquid units selected; Test type: Superiority; p = 0.076, Mixed Models Analysis

3. Secondary Outcome: Motivation to Quit Smoking Cigarettes
Description: Based on a question asking how motivated from 1 (not at all) to 10 (extremely) the participant is to quit smoking cigarettes at this time
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Menthol Ban Only for Cigarettes | Menthol Ban for Cigarettes and E-cigarettes | No Menthol Ban
Number analyzed (Participants) | 16 | 15 | 16
units on a scale | 3.6 (2.2) | 3.1 (2.2) | 3.2 (1.7)
Statistical Analysis 1: Comparison: Menthol Ban Only for Cigarettes vs Menthol Ban for Cigarettes and E-cigarettes vs No Menthol Ban; Test type: Superiority; p = 0.27, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: For the duration of each participant's participation (up to 6 weeks for each participant)
Description: Adverse events rated as possibly, probably or definitely related to being in the study
Arm/Group | Menthol Ban Only for Cigarettes | Menthol Ban for Cigarettes and E-cigarettes | No Menthol Ban
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 2/15 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Menthol Ban Only for Cigarettes (N=16) | Menthol Ban for Cigarettes and E-cigarettes (N=15) | No Menthol Ban (N=16)
throat irritation / cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
pain / discomfort during inhalation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03402243/Prot_SAP_000.pdf